CLINICAL TRIAL: NCT02649413
Title: Adjusted Steroid Therapy in Children With Idiopathic Nephrotic Syndrome
Brief Title: Adjusted Steroids Therapy in Childerens With Idiopathic Nephrotic Syndrome
Acronym: AJSNS
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Rabin Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 695 RMC -AJSNS
Record Dates: First submitted 2015-12-31; First posted 2016-01-07 (Estimated); Last update posted 2016-01-12 (Estimated); Status verified 2015-12

CONDITIONS: Nephrotic Syndrome, Minimal Change
MeSH Terms: conditions — Nephrosis, Lipoid | interventions — Prednisone; Adrenal Cortex Hormones

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Early response to prednisone treatment (Experimental): intervention -children that will have a remission in 8 days (response) will get an adjusted steroids dose treatment.children that have a remission between 9-28 days will get a regular steroid dose.
  Interventions: Drug: Prednisone

INTERVENTIONS:
Drug: Prednisone — Children with Idiopathic Nephrotic syndrome will start 60 mg/m2 prednisone.children that response in 8 days will receive an adjusted dose while the rest of the group will receive the 4 weeks usually dose.
  Other Names: corticosteroids

SUMMARY:
The initial steroids dose for Nephrotic Syndrome is 60mg/1m2 for 6-4 weeks and the duration of the first steroid course is between 8 weeks to 6 months. The base of the initial dose for steroids Idiopathic nephrotic syndrome been put in the early 70s. In our study the investigators will adjusted the first steroids does to the response day. Our primary end point is : a lower adjusted dose is as good as the fix dose in the first year after diagnosis.

DETAILED DESCRIPTION:
About 90% of the patients will response to steroid therapy. The initial steroid dose is between 2mg/kg or 60mg/1m2 for 6-4 weeks and the duration of the first steroid course is between 8 weeks to 6 months. The bases of this treatment have been put in the early 70s. Since then most of the study were focused on the duration of the therapy with a results that 8-12 weeks course is as good as 6 month. Studies have showed no difference in response rate between 2mg/kg to 60m2' although the difference in the dose in young children can rich to 25%. Other retrospective analysis been show that patients who response in the first 7-9 days tend to have lass relapses than other patients. In our nephrology clinic the investigators there is ongoing clinical study on low doses of steroid therapy for relapse of nephritic syndrome with good results.

ELIGIBILITY:
Inclusion Criteria:

* Children who recently have been diagnosed with nephrotic syndrome.

Exclusion Criteria:

* Children with nephrotic syndrome that can not be treated with steroids.

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 75 (Estimated)
Dates: Start 2016-03; Primary Completion 2019-04 (Estimated); Study Completion 2019-06 (Estimated)

PRIMARY OUTCOMES:
The time until the first relapse | 6 months
  All Children with Nephrotic Syndrome will start a dose of 60 mg/m2 prednisone.patients that will response in 8 days (the first day with a negative or trace in the urine deep stick test)will receive adjusted lower steroid dose.the outcome is the time until the first relapse( positive protein in deep stick urine test,or low serum albumin with positive urine deep stick).the control group is the historical data from a prospective malty center observation study.

SECONDARY OUTCOMES:
Number of relapse during first year | one year
  We will count the number of relapse episodes in the first year since diagnosis.

CONTACTS AND LOCATIONS:
Overall Officials: Amit Dagan, Dr., Principal Investigator — Shneider children Hospital Nephrology Institute
Locations (1):
- Shneider children Hospital Nephrology Institute, Petah Tikva, Israel

IPD SHARING:
Plan to Share IPD: No